CLINICAL TRIAL: NCT04937023
Title: Assessing the Clinical Efficacy of Ursodeoxycholic Acid (Udca) as a Local Drug Delivery Agent in the Treatment of Intra-bony Defects: A Clinico-radiographic Study
Brief Title: Ursodeoxycholic Acid (Udca) as a Local Drug Delivery Agent in the Treatment of Intra-bony Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/1/2020
Record Dates: First submitted 2021-06-17; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Bone Regeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UDCA gel will be injected using a syringe with blunt cannula into the defect site (Experimental): In the test group, the prepared UDCA gel will be injected using a syringe with blunt cannula into the two or three wall intra-bony defects with probing pocket depth ≥3mm after performing SRP.
  Interventions: Drug: Ursodeoxycholic acid gel
- placebo gel will be injected in to the defect site using a syringe with blunt cannula. (Placebo Comparator): In patients allocated to control group, placebo gel will be injected in to the defect site using a syringe with blunt cannula after scaling and root planing.
  Interventions: Drug: Ursodeoxycholic acid gel

INTERVENTIONS:
Drug: Ursodeoxycholic acid gel — Following scaling and root planing in intrabony defects UDCA gel will be injected
  Other Names: experimental group

SUMMARY:
The aim of this study is to evaluate the efficacy of ursodeoxycholic acid as local drug delivery agent in intra- bony defect to achieve bone regeneration.

DETAILED DESCRIPTION:
Experimental: Main treatment group the prepared UDCA gel will be injected using a syringe with blunt cannula into the defect site.

Comparator: In patients allocated to control group, placebo gel will be injected in to the defect site using a syringe with blunt cannula.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male and female patients of age>18 years with intrabony defects - two wall or three wall defects and probing pocket depths (PPD) of >3mm will be included

Exclusion Criteria:

* Medically compromised patients, pregnant women, heavy smokers, and patients who underwent radiotherapy or chemotherapy will be excluded.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of bone regeneration | Baseline to 6 months
  Radiovisiography (RVG) will be used to assess bone regeneration achieved post-operatively after 3 months and 6 months.
Evaluation if clinical attachment level | Baseline to 6 months
  Assessment of clinical attachment level (CAL) using UNC-15 probe at baseline and post-operatively at 3 and 6 months.
Evaluation of probing pocket depth | Baseline to 6 months
  Assessment of probing pocket (PPD) depth using UNC- 15 probe at baseline and postoperatively at 3 and 6 months.

SECONDARY OUTCOMES:
Evaluation of gingiva | Baseline to 6 months
  Gingival index (GI) - according to Loe H and Silness P, 1963
Evaluation of gingival bleeding | Baseline to 6 months
  Gingival bleeding index - Ainamo and Bay, 1975

CONTACTS AND LOCATIONS:
Locations (1):
- SVS Institute of Dental Sciences, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No